CLINICAL TRIAL: NCT02844465
Title: Stereotactic Laser Ablation for Temporal Lobe Epilepsy
Brief Title: Stereotactic Laser Ablation for Temporal Lobe Epilepsy (Slate)
Acronym: SLATE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MedtronicNeuro (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS-05000
Record Dates: First submitted 2016-07-15; First posted 2016-07-26 (Estimated); Results first posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Temporal Lobe Epilepsy
Keywords: epilepsy; laser ablation; Visualase; laser interstitial thermal therapy
MeSH Terms: conditions — Epilepsy, Temporal Lobe; Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Treatment (Experimental): Visualase MRI-guided laser ablation procedure
  Interventions: Device: Visualase MRI-Guided Laser Ablation

INTERVENTIONS:
Device: Visualase MRI-Guided Laser Ablation — All subjects will undergo MRI-guided laser ablation of the amygdala and hippocampus with the Visualase System.
  Other Names: Visualase System; Visualase procedure; Laser interstitial thermal therapy; Stereotactic laser ablation

SUMMARY:
The study is designed to evaluate the safety and efficacy of the Visualase MRI-guided laser ablation system for mesial temporal epilepsy (MTLE).

DETAILED DESCRIPTION:
The purpose of the study is to evaluate the safety and efficacy of the Visualase MRI-guided laser ablation system for necrotization or coagulation of epileptogenic foci in patients with intractable mesial temporal lobe epilepsy.

The study will include approximately 150 adult patients with drug-resistant MTLE treated at selected epilepsy centers across the United States. After the Visualase procedure, patients will be followed for 12 months and evaluated for freedom from seizures, quality of life, adverse events, and neuropsychological outcomes.

ELIGIBILITY:
Inclusion Criteria:

* History of drug-resistant mesial temporal lobe epilepsy (MTLE)
* If the subject has a vagus nerve stimulator (VNS), must have failed to achieve sustained seizure freedom with the VNS implanted for at least 6 months
* On stable antiepileptic drugs (AEDs) (and/or stable VNS setting, if applicable) and compliant with medication use
* An average of at least 1 complex partial or secondarily generalized seizure compatible with MTLE per month
* Seizure symptoms and/or auras compatible with MTLE
* Video EEG shows evidence of seizures from one temporal lobe consistent with MTLE
* MRI has evidence consistent with mesial temporal lobe sclerosis
* Willing and able to remain on stable AEDs (and stable VNS setting, if applicable) for 12 months following the Visualase procedure
* Willing and able to comply with protocol requirements
* Able to complete study assessments in English or Spanish language

Exclusion Criteria:

* Unwilling or unable to sign the study informed consent form
* Pregnant or intends to become pregnant during the course of the study
* Currently implanted with a device contraindicating MRI
* Progressive brain lesions and/or tumors not associated with epileptic disease state
* History of previous intracranial surgery for treatment of epileptic seizures
* Persistent extra-temporal or predominant contralateral focal interictal spikes or slowing, or generalized interictal spikes on EEG
* Seizures with contralateral or extra-temporal ictal onset on EEG
* Aura and/or ictal behavior suggest an extra-temporal focus
* MRI evidence of epileptogenic, extra-temporal lesions, dual pathology in the temporal lobe, or contralateral hippocampal MRI increased signal and/or loss of architecture
* If additional testing has been performed, results are discordant with the seizure focus scheduled for ablation
* Non-compliance with AED requirements
* IQ < 70
* Dementia or other progressive neurological disease
* Unstable major psychiatric illness, psychogenic non-epileptic seizures, or medical illness that would contraindicate the Visualase procedure or affect the neuropsychological assessments
* Participation in other research that may potentially interfere with SLATE endpoint(s)
* Allergy to gadolinium

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2023-12-11 (Actual); Study Completion 2023-12-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Gross, MD, PhD, Principal Investigator — Emory University; Michael Sperling, MD, Principal Investigator — Thomas Jefferson University
Locations (23):
- United States (23):
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Stanford University, Palo Alto, California
  - University of California, San Francisco, San Francisco, California
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - University of Miami, Miami, Florida
  - Emory University, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of Louisville Hospital, Louisville, Kentucky
  - Johns Hopkins University, Baltimore, Maryland
  - Henry Ford Health System, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Rutgers University - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Northwell Health, Great Neck, New York
  - Columbia University Medical Center, New York, New York
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - Ohio Health Research Institute, Columbus, Ohio
  - Oregon Health & University Science, Portland, Oregon
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - University of Virginia, Charlottesville, Virginia
  - University of Washington Harborview, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No
There is not a plan to share individual participant data, but aggregate data for all primary and secondary endpoints will be shared.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment
Started | 167
Completed | 107
Not Completed | 60
Not completed — Screen Failure | 36
Not completed — Withdrawal Prior to Procedure | 17
Not completed — Withdrawal by Subject | 5
Not completed — Lost to Follow-up | 1
Not completed — Retreatment | 1

BASELINE CHARACTERISTICS:
Population: Participants who received the Visualase procedure
Arm/Group | Treatment
Number analyzed (Participants) | 114
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.2 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67
  Male | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20
  Not Hispanic or Latino | 94
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 12
  White | 93
  More than one race | 0
  Unknown or Not Reported | 5
Region of Enrollment [Number; unit: participants]
  United States | 114
BMI [Mean (Standard Deviation); unit: kg/m^2] | 27.49 (5.88)
Epilepsy Diagnosis (years from diagnosis) [Mean (Standard Deviation); unit: years] | 24.0 (17.2)
Average Monthly Seizure Frequency over the 12 Months Prior to Enrollment: All Seizure Types [Mean (Standard Deviation); unit: seizures] | 11.5 (15.4)
Language Dominance [Count of Participants; unit: Participants]
  Left | 53
  Right | 6
  Bilateral | 4
  Inconclusive | 1
  Not Evaluated | 50
Subject Handedness [Count of Participants; unit: Participants]
  Left-handed | 15
  Right-handed | 97
  Mixed-handed | 2
Vague Nerve Stimulator Currently Implanted [Count of Participants; unit: Participants] | 5
Side of Brain Intended for MRI-Guided Stereotactic Laser Ablation [Count of Participants; unit: Participants]
  Left | 74
  Right | 40

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Qualifying Adverse Events
Description: The incidence of qualifying device, procedure and/or anesthesia related adverse events. These events must also be moderate or severe and permanent for the following AEs: anxiety, aphasia, blurry vision, depression, diplopia, emotional lability, hemianopia, hemiparesis, memory impairment/difficulty, neurologic deficits, paralysis, psychological/psychiatric complications, quadrantanopia, sensory loss, sleep problems or insomnia. An exact 95% confidence interval (CI) will be calculated to determine if the upper bound of the CI for qualified AEs is less than 40%.
Time Frame: 12 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment
Number analyzed (Participants) | 114
percentage of participants | 7.9 [3.7 to 14.5]

2. Primary Outcome: Seizure Freedom, Defined as Engel Classification of Postoperative Outcome Class I
Description: Seizure freedom at 12 months following the Visualase procedure (starting at 30 days post-procedure through 365 days post procedure). Engel Class I: Free of disabling seizures includes subclasses: A. Completely seizure free since surgery, B. Nondisabling simple partial seizures only since surgery, D. Generalized convulsions with antiepileptic drugs (AED) discontinuation only. An exact 95% CI will be calculated to determine if the lower bound of the CI for seizure freedom at 12 months following the Visualase procedure will be greater than 43%. Multiple imputation was used if subject diary data was not compliant. Retreated subjects are treated as failures.
Time Frame: 12 months
Measure: Number (95% Confidence Interval); unit: percentage of subjects Engel Class I
Arm/Group | Treatment
Number analyzed (Participants) | 114
percentage of subjects Engel Class I | 56.0 [46.2 to 65.8]

3. Secondary Outcome: Seizure Freedom Compared to Historical Controls (Medical Therapy)
Description: Seizure freedom (Engel Class I) compared to historical control for continued medical therapy. It is hypothesized that the seizure freedom at 12 months following the Visualase procedure will be superior to 8% reported in the literature for continued medical therapy. An exact 95% CI for the percentage of subjects who are seizure free will be calculated.
Time Frame: 12 months
Measure: Number (95% Confidence Interval); unit: percentage of subjects Engel Class I
Arm/Group | Treatment
Number analyzed (Participants) | 114
percentage of subjects Engel Class I | 56.0 [46.2 to 65.8]

4. Secondary Outcome: Seizure Freedom, Including Subjects Retreated With Visualase
Description: Seizure freedom (Engel Class I) including subjects who were retreated with Visualase. The outcome after retreatment will count towards the endpoint. It is hypothesized that the lower bound of the 95% CI for seizure freedom at 12 months following the Visualase procedure, including subjects retreated with Visualase, will be greater than 43%. Subjects retreated with Visualase will count toward the secondary efficacy endpoint based on their outcome after retreatment. If they have become seizure free and have reached 12 months follow-up from time of retreatment, they are counted as seizure free. Otherwise, they will count as not seizure free. An exact 95% CI will be calculated to determine if the lower bound of the CI for seizure freedom at 12 months following a subject's last Visualase procedure, including patients retreated with Visualase, will be greater than 43%.
Time Frame: 12 months
Measure: Number (95% Confidence Interval); unit: percentage of subjects Engel Class I
Arm/Group | Treatment
Number analyzed (Participants) | 114
percentage of subjects Engel Class I | 56.0 [46.2 to 65.8]

5. Secondary Outcome: Change in Boston Naming Test Scores
Description: Within-subject change of Boston Naming Test score (English language version) from baseline to 12 months following the Visualase procedure. The Boston Naming Test is a neuropsychological assessment tool to measure confrontational word retrieval. The test contains 60 line drawings graded in difficulty which the participants need to name. The total score ranges from 0-60 with a higher score meaning a better outcome.
Time Frame: Baseline and 12 months
Population: Participants who had both a baseline and 12 month BNT total score
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 89
score on a scale | -0.1 (7.2)
Statistical Analysis 1: Comparison: Treatment; It is hypothesized that the Boston Naming Test score will not decrease from baseline to 12 months following the Visualase procedure. The hypotheses associated with this endpoint are as follows: Null Hypothesis: μ (V-BNT - BSL-BNT) + δ ≤ 0 Alternate Hypothesis: μ (V-BNT - BSL-BNT) + δ > 0 Where μ (V-BNT - BSL-BNT) = mean difference in the Boston Naming Test score from baseline to Month 12 post Visualase; Test type: Non-Inferiority — A non-inferiority test will be performed using a paired t-test, with a non-inferiority delta (δ) of one Reliable Change Index (RCI) of 5 points, to test the hypothesis of no reduction. A two-tailed alpha of 0.05 will be used; p < 0.0001, Paired t-test

6. Secondary Outcome: Change in Rey Auditory Verbal Learning Test Scores
Description: Within-subject change of Rey Auditory Verbal Learning Test (RAVLT) 5-Trial Total score (English language version) from baseline to 12 months following the Visualase procedure. It is used for assessing episodic memory by providing scores for evaluating different aspects of memory. The RAVLT presents a list of 15 words across 5 consecutive trials. The list is read to the participant and the participant is asked to recall as many words as possible. This is repeated for 5 consecutive trials. The scores range from 0-75 with a higher score indicating a better outcome.
Time Frame: Baseline and 12 months
Population: Participants with both a baseline and 12 month RAVLT 5-Trial Total Learning Score
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 92
score on a scale | -0.9 (8.9)
Statistical Analysis 1: Comparison: Treatment; It is hypothesized that the Rey Auditory Verbal Learning Test 5-Trial Total score will not decrease from baseline to 12 months following the Visualase procedure. The hypotheses associated with this endpoint are as follows: Null Hypothesis: μ (V-RAVLT - BSL-RAVLT) + δ ≤ 0 Alternate Hypothesis: μ (V-RAVLT - BSL-RAVLT) + δ > 0 Where μ (V-RAVLT - BSL-RAVLT) = mean difference in the Rey Auditory Verbal Learning Test 5-Trial Total score from baseline to Month 12 post Visualase; Test type: Non-Inferiority — A non-inferiority test will be performed using a paired t-test, with a non-inferiority delta (δ) of one Reliable Change Index (RCI) of 15 points, to test the hypothesis of no reduction. A two-tailed alpha of 0.05 will be used; p < 0.0001, Paired t-test

7. Secondary Outcome: Change in Quality of Life in Epilepsy (QOLIE-31) Scores
Description: Within-subject change of the QOLIE-31 score (English language version) from baseline to 12 months following the Visualase procedure, categorized as -1 if the decrease is clinically significant (<= -11.8), categorized as 0 if not clinically significant (-11.7 to +11.7), and categorized as +1 if the increase is clinically significant (>= 11.8). The QOLIE-31 evaluates a participant's quality of life in relation to their epilepsy. It is used to asses a person's overall wellness, including their social functioning and cognitive impact. The QOLIE scores range from 0-100 with a higher score meaning a better outcome.
Time Frame: Baseline and 12 months
Population: Participants who had both a baseline and 12 month QOLIE English language version assessment completed
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 93
Participants
  Clinically Significant Decrease (<=-11.8) | 1
  Non-Clinically Significant Change (-11.7 to +11.7) | 54
  Clinically Significant Increase (>= 11.8) | 38
Statistical Analysis 1: Comparison: Treatment; It is hypothesized that the QOLIE-31 score will increase (improve) from baseline to 12 months following the Visualase procedure. The hypotheses associated with this endpoint are as follows: Null Hypothesis: M (V-QOLIE-31 - BSL-QOLIE-31) ≤ 0 Alternate Hypothesis: M (V-QOLIE-31 - BSL-QOLIE-31) > 0 Where M (V-QOLIE-31 - BSL-QOLIE-31) = sign-test statistic ([increases-decreases]/2) in the Quality of Life in Epilepsy inventory from baseline to Month 12 post Visualase; Test type: Other — A sign test will be used to determine if the median categorical change is significantly greater than zero; p < 0.0001, Sign test

8. Secondary Outcome: Change in SF-36 Mental Component Score
Description: Within-subject change of short form (SF)-36 quality of life questionnaire Mental Component Score (English language version) from baseline to 12 month following the Visualase procedure, categorized as -1 if the decrease is clinically significant (<=-4.58), categorized as 0 if not clinically significant (-4.57 to +4.57), and categorized as +1 if the increase is clinically significant (>=4.58). The SF-36 is a 36-item, patient-reported survey of patient health. It consists of eight scaled scores, which are the weighted sums of the questions in their section. The SF-36 Mental Component Score ranges from 0-100 with a higher score meaning a better outcome, on the assumption that each questions carries equal weight.
Time Frame: Baseline and 12 Months
Population: Number of participants who had both a baseline and 12 month Mental Component Score in English.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 85
Participants
  Clinically Significant Decrease (<= - 4.58) | 13
  Non-Clinically Significant Change (-4.57 to +4.57) | 33
  Clinically Significant Increase (>=4.58) | 39
Statistical Analysis 1: Comparison: Treatment; It is hypothesized that the SF-36 Mental Component Score (MCS) will increase (improve) from baseline to 12 months following the Visualase procedure. The hypotheses associated with this endpoint are as follows: Null Hypothesis: M (V-SF-36 - BSL-SF-36-MCS) ≤ 0 Alternate Hypothesis: M (V-SF-36 - BSL-SF-36-MCS) > 0 Where M (V- SF-36-MCS - BSL- SF-36-MCS) = sign-test statistic ([increases-decreases]/2) in the SF-36 quality of life questionnaire MCS from baseline to Month 12 post Visualase; Test type: Other — A sign test will be used to determine if the median categorical change is significantly greater than zero; p = 0.0004, Sign test

9. Secondary Outcome: Change in SF-36 Physical Component Score
Description: Within-subject change of short form (SF)-36 quality of life questionnaire Physical Component Score (English language version) from baseline to 12 month following the Visualase procedure, categorized as -1 if the decrease is clinically significant (<=-3.02), categorized as 0 if not clinically significant (-3.01 to +3.01), and categorized as +1 if the increase is clinically significant (>=3.02). The SF-36 is a 36-item, patient-reported survey of patient health. It consists of eight scaled scores, which are the weighted sums of the questions in their section. The SF-36 Physical Component Scores range from 0-100 with a higher score meaning a better outcome, on the assumption that each questions carries equal weight.
Time Frame: Baseline and 12 Months
Population: Participants who had both a baseline and 12 month SF-36 Physical Component Score in English.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 84
Participants
  Clinically Significant Decrease (<=-3.02) | 12
  Non-Clinically Significant Change (-3.01 to +3.01) | 28
  Clinically Significant Increase (>= 3.02) | 44
Statistical Analysis 1: Comparison: Treatment; It's hypothesized that the SF-36 Physical Component Score (PCS) will increase (improve) from baseline to 12 months following the Visualase procedure. The hypotheses associated with this endpoint are as follows: Null Hypothesis: M (V-SF-36-PCS - BSL-SF-36-PCS) ≤ 0 Alternate Hypothesis: M (V-SF-36-PCS - BSL-SF-36-PCS) > 0 Where M (V-SF-36-PCS - BSL- SF-36-PCS) = sign-test statistic ([increases-decreases]/2) in the SF-36 quality of life questionnaire PCS from baseline to Month 12 post Visualase; Test type: Other — A sign test will be used to determine if the median categorical change is significantly greater than zero; p < 0.0001, Sign test

10. Secondary Outcome: Seizure Freedom Compared to Historical Controls (Open Surgical Resection)
Description: Seizure freedom (Engel Class I) compared to historical control for open surgical resection.
  It is hypothesized that the seizure freedom at 12 months following the Visualase procedure will not be inferior to 64% reported in the literature for open surgical resection.
  An exact 95% CI for the percentage of subjects who are seizure free will be calculated and its lower boundary compared to zero after subtraction of the historical open surgical resection percentage of 64% and the addition of the equivalence delta percentage of 10%.
Time Frame: 12 Months
Measure: Number (95% Confidence Interval); unit: percentage of subjects Engel Class I
Arm/Group | Treatment
Number analyzed (Participants) | 114
percentage of subjects Engel Class I | 56.0 [46.2 to 65.8]
Statistical Analysis 1: Comparison: Treatment; Test type: Non-Inferiority — The hypotheses associated with this endpoint are: Null Hypothesis: π V - 64% + δ ≤ 0 Alternate Hypothesis: π V - 64% + δ > 0 Where πV is the proportion of subjects treated with Visualase experiencing no seizures. An exact 95% CI for the percentage of subjects who are seizure free will be calculated and its lower boundary compared to zero after subtraction of the historical open surgical resection percentage of 64% and the addition of the equivalence delta percentage of 10%; Proportion of Participants = 56.0, 95% CI 2-sided [46.2 to 65.8]

ADVERSE EVENTS:
Time Frame: Enrollment to 12 months post procedure
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 0/167
Serious Adverse Events (participants affected / at risk) | 16/167
Other Adverse Events (participants affected / at risk) | 31/167
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=167)
Pharyngitis (Infections and infestations) | 1 (1)
Postoperative wound infection (Infections and infestations) | 1 (1)
Meningitis chemical (Injury, poisoning and procedural complications) | 1 (1)
Blood sodium decreased (Investigations) | 1 (1)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Focal dyscognitive seizures (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 1 (1)
Memory impairment (Nervous system disorders) | 1 (1)
Partial seizures with secondary generalisation (Nervous system disorders) | 1 (1)
Psychogenic seizure (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Status epilepticus (Nervous system disorders) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1)
Mental status changes (Psychiatric disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=167)
Headache (Nervous system disorders) | 13 (13)
Quadrantanopia (Nervous system disorders) | 21 (21)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PIs are required to submit proposals through the publication committee and receive approval from the publication committee before publishing results.

DOCUMENTS (2):
  • Study Protocol (2018-04-09): https://cdn.clinicaltrials.gov/large-docs/65/NCT02844465/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-01): https://cdn.clinicaltrials.gov/large-docs/65/NCT02844465/SAP_001.pdf